CLINICAL TRIAL: NCT06506292
Title: A Phase II Trial of Perioperative Adebrelimab Combined With XELOX in Resectable Locally Advanced Gastric/Gastroesophageal Junction Cancer (GC/GEJC)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202407-GC/GEJC
Record Dates: First submitted 2024-07-11; First posted 2024-07-17 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Adebrelimab (SHR-1316); XELOX; GC/GEJC
MeSH Terms: interventions — XELOX

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study arm (Experimental): Neoadjuvant therapy:
  Adebrelimab: 1200 mg, iv, d1, q3w, 3 cycles of treatment; XELOX regimen: oxaliplatin: 130 mg/m2,iv,d1; capecitabine: 1000 mg/m2,po,pid,d1-d14; q3w, 3 cycles;
  Surgery within 3-6 weeks of the end of neoadjuvant therapy, with adjuvant therapy starting 4-6 weeks after surgery.
  Postoperative adjuvant therapy： Adebrelimab: 1200 mg, iv, d1; q3w, 5 cycles of treatment; XELOX regimen: oxaliplatin: 130 mg/m2,iv,d1; capecitabine: 1000 mg/m2,po,pid,d1-d14; q3w, treatment for 5 cycles;
  Perioperative adebelizumab combined with XELOX chemotherapy for a total of no more than 8 cycles of treatment.
  Maintenance therapy:
  Adebrelimab maintenance therapy up to 1 year.
  Interventions: Drug: Adebrelimab; Drug: XELOX

INTERVENTIONS:
Drug: Adebrelimab — Adebrelimab:1200 mg, iv, d1
Drug: XELOX — oxaliplatin: 130 mg/m2,iv,d1; capecitabine: 1000 mg/m2,po,pid,d1-d14

SUMMARY:
To observe and evaluate the efficacy and safety of adebrelimab combination chemotherapy regimen in the perioperative treatment of surgically resectable gastric cancer/adenocarcinoma of the gastroesophageal junction.

DETAILED DESCRIPTION:
Gastric cancer is the fifth most common cancer in the world and ranks fourth in mortality. Radical surgery is the main treatment for resectable gastric cancer. For patients with progressive gastric cancer, especially those with stage IIIB and IIIC, their 5-year overall survival (OS) rate after radical surgery is still difficult to exceed 50%. Although D2 radical surgery and postoperative adjuvant chemotherapy have significantly improved the prognosis of patients with progressive gastric cancer, the recurrence rate is still as high as 50%~80%. Several therapeutic approaches have been established to reduce the risk of recurrence and improve long-term survival, including perioperative chemotherapy, adjuvant chemotherapy, and adjuvant radiotherapy. The effect of adding targeted therapies and/or immune checkpoint inhibitors (ICIs) to neoadjuvant/adjuvant therapies is currently being studied. While multiple programmed death 1 (PD-1) inhibitors have been approved for first/third line treatment of unresectable/metastatic gastric cancer. However, the role of immune checkpoint inhibitors in resectable gastric cancer remains unclear and is being investigated in various clinical trials.

We conducted this study with 8 cycles of perioperative treatment with adebrelimab in combination with XELOX chemotherapy regimen and adebelizumab maintenance therapy up to 1 year. To observe and evaluate the efficacy and safety of adebrelimab combination chemotherapy regimen in the perioperative treatment of surgically resectable gastric cancer/adenocarcinoma of the gastroesophageal junction.

ELIGIBILITY:
Inclusion Criteria:

1. Patients voluntarily enrolled in the study and signed an informed consent form
2. 18-75 years old, male and female gender are not limited
3. Gastric adenocarcinoma or adenocarcinoma of the gastroesophageal junction as determined by pathologic histology
4. Clinical staging of II-III/T3-4aNxM0 (AJCC 8th edition cTNM staging of gastric cancer)
5. Clinically judged to be surgically resectable
6. have at least one measurable lesion (according to the requirements of RECISTv1.1, the long diameter of spiral CT scan of this measurable lesion is ≥10mm or the short diameter of enlarged lymph node is ≥15mm)
7. No other anti-tumor therapy has been received
8. ECOG score:0~1
9. Good function of major organs
10. No active hepatitis B virus (HBV) infection
11. Women of childbearing potential must have had a negative blood pregnancy test within 3 days prior to randomization and be willing to use an appropriate method of contraception during the trial and for 6 months after completion of treatment. For men, surgical sterilization or agreement to use an appropriate method of contraception during the study and for 3 months after completion of treatment.

Exclusion Criteria:

1. patients who are pregnant or breastfeeding
2. Received prior anti-tumor therapy, including chemotherapy, radiotherapy, targeted therapy, or immunotherapy
3. other malignant tumor (except basal or squamous cell carcinoma, superficial bladder cancer, cervical cancer in situ or breast cancer) within the past 5 years
4. Uncontrolled pleural effusion, pericardial effusion or ascites
5. Clinically determined to be inoperable or with distal metastasis
6. Severe cardiovascular disease, such as symptomatic coronary artery disease, class ≥II congestive heart failure, uncontrolled arrhythmia, myocardial infarction, within 12 months prior to enrollment.
7. Complicated upper gastrointestinal tract obstruction/bleeding or digestive dysfunction or malabsorption syndrome
8. History of gastrointestinal perforation in the 6 months prior to enrollment
9. Severe uncontrolled co-infection or other severe uncontrolled concomitant disease, moderate or severe renal impairment
10. Have clinical symptoms or diseases of the heart that are not well controlled, such as: (1) Grade II or higher cardiac insufficiency according to the New York Heart Association (NYHA) criteria (see Appendix 5) or cardiac ultrasound: LVEF (Left Ventricular Ejection Fraction) < 50%; (2) Unstable angina pectoris; (3) Myocardial infarction within 1 year prior to the initiation of study treatment; (4) Clinically significant supraventricular or ventricular arrhythmia requiring treatment or intervention; (5) QTc>450ms (men); QTc>470ms (women) (QTc interval calculated by the Fridericia formula; in case of QTc abnormality, three consecutive measurements can be taken at 2-minute intervals and averaged)
11. have an allergic reaction to the drugs used in the study
12. Use of immunosuppressive drugs within 4 weeks prior to the first dose of study treatment, excluding topical glucocorticosteroids by nasal, inhalational, or other routes or physiologic doses of systemic glucocorticosteroids (i.e., no more than 10 mg/day of prednisone or equivalent doses of other glucocorticosteroids), or use of hormones for the prevention of contrast allergy
13. known history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation
14. current concomitant interstitial pneumonitis or interstitial lung disease, or a prior history of interstitial pneumonitis or interstitial lung disease requiring hormonal therapy, or other conditions that may interfere with the determination and management of immune-related pulmonary toxicity such as pulmonary fibrosis, mechanized pneumonitis (e.g., occlusive bronchiectasis), pneumonias, drug-associated pneumonias, idiopathic pneumonias, or active pneumonitis as seen on screening chest computed tomography (CT) maps Evidence of or severely impaired lung function in subjects with a history of radiation pneumonitis in the permitted radiation field, active tuberculosis
15. presence of active autoimmune disease or history of autoimmune disease with potential for relapse (including, but not limited to: autoimmune hepatitis, interstitial pneumonitis, uveitis, enteritis, pituitary gland inflammation, vasculitis, nephritis, hyperthyroidism, and hypothyroidism [subjects who can be controlled by hormone replacement therapy only are eligible for enrollment]); subjects with a dermatological condition that does not require systemic treatment such as vitiligo psoriasis, alopecia areata, controlled type I diabetes mellitus treated with insulin or asthma that has completely resolved in childhood and does not require any intervention in adulthood may be included; asthmatics requiring medical intervention with bronchodilators may not be included
16. Immunosuppressive or systemic hormone therapy for immunosuppression within 14 days prior to initiation of study treatment (doses >10 mg/day of prednisone or other equipotent hormone)
17. severe infection within 4 weeks prior to initiation of study treatment, including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia; therapeutic antibiotics given orally or intravenously within 2 weeks prior to initiation of study treatment (patients receiving prophylactic antibiotics (e.g., for prevention of urinary tract infection or exacerbation of COPD are eligible for study participation))
18. Patients with congenital or acquired immune deficiency (e.g., HIV-infected)
19. Use of immunosuppressive medications within 4 weeks prior to the first dose of study drug
20. live attenuated vaccine within 4 weeks prior to the first dose or plan to receive live attenuated vaccine during the study period
21. previous treatment with other anti-PD-1 antibodies or other immunotherapy against PD-1/PD-L1;
22. permitted palliative radiotherapy to non-target lesions for symptom control, which must have been completed at least 2 weeks prior to initiation of study treatment use, with no recovery from radiotherapy-induced adverse events to ≤ CTCAE grade 1
23. received other experimental drug therapy within 28 days prior to initiation of study treatment
24. In the judgment of the investigator, the patient has other factors that may affect the results of the study or cause this study to be forced to be terminated in midstream, such as alcoholism, drug abuse, other serious illnesses (including psychiatric illnesses) that require comorbid treatment, serious laboratory test abnormalities, accompanied by family or social factors that would affect the patient's safety.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Pathological completeresponse, pCR | After surgical excision with follow up of an average of 1 year
  Disappearance of tumor cells from resected specimen

SECONDARY OUTCOMES:
Major Pathological response, MPR | After surgical excision with follow up of an average of 1 year
  the percentage of tumor cells before and after treatment was compared according to biopsy specimens before neoadjuvant therapy and pathological specimens after surgery; the percentage of tumor cells was evaluated on resected tumor slides. MPR was defined as ≤ 10% tumor cells.
Objective response rate,ORR | From treatment initiation to progressive disease or EOT due to any cause, assessed up to 1 year
  Defined as proportion of patients who have a best response of CR or PR
R0 resection rate | After surgical excision with follow up of an average of 1 year
  Patients who underwent radical resection as a percentage of the total number of patients who underwent surgical resection
Event Free Survival, EFS | From treatment initiation to progressive disease, discontinuation of the treatment for any reason, or death due to any cause, assessed up to 1 year
  From date of surgery until the date of recurrence detection.
Disease control rate, DCR | From treatment initiation to progressive disease or EOT due to any cause, assessed up to 1 year
  Defined as proportion of patients who have CR or PR or SD
Disease-free survival, DFS | From treatment initiation to cancer recurrence or death due to any cause, assessed up to 1 year
  Duration of survival before cancer recurrence or death
Overall Survival, OS | From treatment initiation until death due to any cause, assessed up to 3 year
  Defined as the time from enrollment to death from any cause
AE/SAE | Up to 1 year
  Incidence of Adverse Events (AE)/Serious Adverse Events (SAE) (as measured by NCI-CTCAE 5.0)

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No